CLINICAL TRIAL: NCT00349128
Title: A Randomized, Double-Blind Trial Assessing the Efficacy and Safety of Low and Standard Doses of Fenofibrate in Combination With Metformin on the Lipid Profile in Patients With Type 2 Diabetes and Dyslipidemia.
Brief Title: Fenofibrate in Dyslipidemia and Metformin-Controlled Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C LF23-0121 03 01
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2007-08

CONDITIONS: Dyslipidemia/Glucose Metabolism Disorder
Keywords: Treatment of Dyslipidemia and of Type 2 Diabetes Mellitus
MeSH Terms: conditions — Dyslipidemias; Glucose Metabolism Disorders | interventions — Fenofibrate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: fenofibrate and metformin combination (drug)

SUMMARY:
The primary objective was to assess the effect of 3-month treatment of low and standard doses of fenofibrate in combination with stable dose of metformin on fasting triglycerides levels in patients with type 2 diabetes and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus

Exclusion Criteria:

* Type 1 diabetes, uncontrolled type 2 diabetes, - HbA1c ≥ 10 % - Fasting plasma glucose > 300 mg/dL - Triglycerides > 500 mg/dL

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382
Dates: Start 2004-01

PRIMARY OUTCOMES:
Change in fasting triglycerides.

SECONDARY OUTCOMES:
Assessment of lipid and glucose metabolisms.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (51):
- Poland (4):
  - Site 201, Katowice
  - Site 203, Katowice
  - Site 202, Warsaw
  - Site 204, Zabrze
- Ukraine (12):
  - Site 111, Dnipropetrovsk
  - Site 113, Dnipropetrovsk
  - Site 108, Kharkiv
  - Site 109, Kharkiv
  - Site 101, Kyiv
  - Site 102, Kyiv
  - Site 103, Kyiv
  - Site 104, Kyiv
  - Site 105, Kyiv
  - Site 106, Kyiv
  - Site 107, Kyiv
  - Site 112, Zaporizhya
- United Kingdom (35):
  - Site 35, Acomb
  - Site 21, Atherstone
  - Site 14, Balsall Common
  - Site 32, Bangor
  - Site 23, Barry
  - Site 36, Basingstoke
  - Site 8, Bexhill-on-Sea
  - Site 20, Camberley
  - Site 22, Chesterfield
  - Site 10, Chippenham
  - Site 13, Coventry
  - Site 31, Doncaster
  - Site 15, Downpatrick
  - Site 17, Ely
  - Site 4, Ely
  - Site 11, Fife
  - Site 1, Frome
  - Site 16, Harrow
  - Site 5, Hastings
  - Site 26, Haverfordwest
  - Site 19, Keresley End
  - Site 9, Kingswood
  - Site 25, Newtownabbey
  - Site 33, Northampton
  - Site 28, Odiham
  - Site 3, Paignton
  - Site 12, Peterborough
  - Site 7, Randalstown
  - Site 27, Slough
  - Site 6, Soham
  - Site 2, South Glamorgan
  - Site 34, Stratford-upon-Avon
  - Site 29, Swindon
  - Site 30, Trowbridge
  - Site 18, Yaxley